CLINICAL TRIAL: NCT02674360
Title: Randomized Controlled Trial Regarding (RCT) Innovative Dissemination Strategies for a Brief Shared Decision Making (SDM) Intervention for Oncologists: Web-based SDM Online Training and Individualized, Context-based Face-to-face SDM Training
Brief Title: RCT Regarding SDM Online Training and Face-to-face SDM Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Heidelberg (Other)
Collaborators: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Principal Investigator, Dr. Kathrin Gschwendtner, Prinicipal Investigator, University Hospital Heidelberg
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: DKH109956, DKH110010
Record Dates: First submitted 2016-01-25; First posted 2016-02-04 (Estimated); Last update posted 2019-06-11 (Actual); Status verified 2019-06

CONDITIONS: Doctor-Patient-Communication

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- SDM Online Training (Active Comparator): The intervention consists of a SDM training for oncologists, which is conducted in the form of a web-based SDM online Training (intervention group I). During training, the oncologists are guided to use decision aids for breast and colon cancer patients in their consultations, which were developed and evaluated in a previous project. The SDM training has the same duration (one session à 120 minutes) in both intervention groups. Doctors in the intervention group receive decision aids for breast cancer and colorectal cancer patients during training. The training contents are based on an already developed, evaluated and published SDM manual. The SDM online training works on the modeling principle.
  Interventions: Behavioral: SDM Training
- Face-to-Face SDM Training (Active Comparator): The intervention consists of a SDM training for oncologists, which is conducted in the form of an individualized, context-based SDM individual face-to-face training at the workplace of the participants (intervention group II). During training, the oncologists are guided to use decision aids for breast and colon cancer patients in their consultations, which were developed and evaluated in a previous project. The SDM training has the same duration (one session à 120 minutes) in both intervention groups. Doctors in the intervention group receive decision aids for breast cancer and colorectal cancer patients during training. The training contents are based on an already developed, evaluated and published SDM manual. The individual training works on the coaching principle.
  Interventions: Behavioral: SDM Training
- Control Group (No Intervention): The Control Group receives no SDM Training. All participants of the Control Group will be offered to participate in the SDM Online Training after T2.

INTERVENTIONS:
Behavioral: SDM Training
  Arms: Face-to-Face SDM Training; SDM Online Training

SUMMARY:
Cancer patients often report that they are not included in important treatment decisions. Numerous studies have shown that a training concerning Shared Decision Making (SDM) for physicians can improve this situation. This does not only lead to a better quality of the doctor-patient interaction, but may have a positive long term impact on treatment adherence, the psychological well-being and the coping abilities of the patients. However, previous experience regarding the implementation of SDM training programs show that it is difficult to recruit physicians for an external SDM group training due to the extensive workload of the physicians. In light of the available evidence on the effectiveness of SDM training and the low motivation by oncologists for traditional SDM group training, this study aims to develop and evaluate a brief SDM intervention. This intervention is disseminated in two different ways which both might be attractive for oncologists. On the one hand an individual face-to-face context-based SDM training is designed and conducted by a trainer at the workplace of the participating oncologists. On the other hand a web-based SDM online training is developed. Both SDM interventions are developed on the basis of an SDM manual evaluated in previous studies.

This study therefore aims to examine the effectiveness of different disseminations strategies (individualized face-to-face context-based SDM individual training vs. web-based SDM online training) compared to a control group without any training. It will be analyzed which improvements in medical SDM competence can be accomplished by the different SDM trainings. Further the effects of the training on SDM knowledge, quality of the doctor-patient interaction and SDM self-efficacy expectation will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Oncologists or physicians treating a significant percentage of breast and/or colorectal cancer patients
2. Internet access

Exclusion Criteria:

* No Exclusion Criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 161 (Actual)
Dates: Start 2016-05; Primary Completion 2018-12-31 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
Change from baseline in SDM competence measured by an objective Rating (OPTION) | T0 (2 weeks before Training) and T1 (1 weeks after Training)
  To measure the SDM competence the OPTION scale (Observing Patient Involvement; Elwyn et al., 2003; Elwyn et al., 2005; Goss et al., 2007.) will be used. The OPTION scale is a validated instrument for measuring the process steps of Shared Decision Making. The consultations are assessed on the basis of 12 items. It shows good reliability with a value of 0.79. The Option rating is based on video recordings and anonymised transcripts. A consultation will be assessed by two blinded raters. The average value per item is used as final value. For the consultations standardized patients are deployed.

SECONDARY OUTCOMES:
Change from baseline in SDM competence by subjective standardized patient rating (Dyadic Option) | T0 (2 weeks before Training), T1 (1 weeks after Training), T2 (3 month after T1)
  Dyadic OPTION (Melbourne et al., 2010), patient version
Change from baseline in SDM competence by subjective standardized patient rating (Patient Perception Scale) | T0 (2 weeks before Training), T1 (1 weeks after Training), T2 (3 month after T1)
  Patient Perception Scale (PPS; Janz et al., 2004)
Change from baseline in SDM competence by subjective standardized patient rating (SDM-Q-9) | T0 (2 weeks before Training), T1 (1 weeks after Training), T2 (3 month after T1)
  SDM-Q-9 (Kriston et al, 2010; Simon, Loh, & Haerter, 2007)
Change from baseline in SDM competence by subjective physician rating (Dyadic Option) | T0 (2 weeks before Training), T1 (1 weeks after Training), T2 (3 month after T1)
  Dyadic OPTION (Melbourne et al., 2010), physician version
Change from baseline in SDM competence by subjective physician rating (Physician-Perception-Scale) | T0 (2 weeks before Training), T1 (1 weeks after Training), T2 (3 month after T1)
  Physician-Perception-Scale (PPS; Janz et al., 2004)
Change from baseline in SDM competence by subjective physician rating (SDM-Q-9) | T0 (2 weeks before Training), T1 (1 weeks after Training), T2 (3 month after T1)
  SDM-Q-Doc (Scholl et al., 2012)
Change from baseline in quality of doctor-patient-interaction by subjective Patient rating (Questionnaire on the Quality of physician-patient interaction) | T0 (2 weeks before Training), T1 (1 weeks after Training), T2 (3 month after T1)
  Questionnaire on the Quality of physician-patient interaction (QQPI, Bieber et al., 2010), Patient version
Change from baseline in quality of doctor-patient-interaction by subjective Physician rating (Questionnaire on the Quality of physician-patient interaction) | T0 (2 weeks before Training), T1 (1 weeks after Training), T2 (3 month after T1)
  Questionnaire on the Quality of physician-patient interaction (QQPI, Bieber et al., 2010), physician version

CONTACTS AND LOCATIONS:
Overall Officials: Christiane Bieber, PD, Principal Investigator — University Hospital Heidelberg
Locations (2):
- Germany (2):
  - University Hospital Heidelberg, Heidelberg, Baden-Wurttemberg
  - University Hospital Hamburg-Eppendorf, Hamburg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Janz NK, Wren PA, Copeland LA, Lowery JC, Goldfarb SL, Wilkins EG. Patient-physician concordance: preferences, perceptions, and factors influencing the breast cancer surgical decision. J Clin Oncol. 2004 Aug 1;22(15):3091-8. doi: 10.1200/JCO.2004.09.069. PMID 15284259
- [Background] Melbourne E, Sinclair K, Durand MA, Legare F, Elwyn G. Developing a dyadic OPTION scale to measure perceptions of shared decision making. Patient Educ Couns. 2010 Feb;78(2):177-83. doi: 10.1016/j.pec.2009.07.009. Epub 2009 Aug 3. PMID 19647970
- [Background] Kriston L, Scholl I, Holzel L, Simon D, Loh A, Harter M. The 9-item Shared Decision Making Questionnaire (SDM-Q-9). Development and psychometric properties in a primary care sample. Patient Educ Couns. 2010 Jul;80(1):94-9. doi: 10.1016/j.pec.2009.09.034. Epub 2009 Oct 30. PMID 19879711
- [Background] Scholl I, Kriston L, Dirmaier J, Buchholz A, Harter M. Development and psychometric properties of the Shared Decision Making Questionnaire--physician version (SDM-Q-Doc). Patient Educ Couns. 2012 Aug;88(2):284-90. doi: 10.1016/j.pec.2012.03.005. Epub 2012 Apr 3. PMID 22480628
- [Background] Bieber C, Muller KG, Nicolai J, Hartmann M, Eich W. How does your doctor talk with you? Preliminary validation of a brief patient self-report questionnaire on the quality of physician-patient interaction. J Clin Psychol Med Settings. 2010 Jun;17(2):125-36. doi: 10.1007/s10880-010-9189-0. PMID 20217195
- [Background] Elwyn G, Edwards A, Wensing M, Hood K, Atwell C, Grol R. Shared decision making: developing the OPTION scale for measuring patient involvement. Qual Saf Health Care. 2003 Apr;12(2):93-9. doi: 10.1136/qhc.12.2.93. PMID 12679504
- [Background] Elwyn G, Hutchings H, Edwards A, Rapport F, Wensing M, Cheung WY, Grol R. The OPTION scale: measuring the extent that clinicians involve patients in decision-making tasks. Health Expect. 2005 Mar;8(1):34-42. doi: 10.1111/j.1369-7625.2004.00311.x. PMID 15713169
- [Background] Goss C, Fontanesi S, Mazzi MA, Del Piccolo L, Rimondini M, Elwyn G, Zimmermann C. Shared decision making: the reliability of the OPTION scale in Italy. Patient Educ Couns. 2007 Jun;66(3):296-302. doi: 10.1016/j.pec.2007.01.002. Epub 2007 Apr 11. PMID 17433603
- [Derived] Muller N, Gschwendtner KM, Dwinger S, Bergelt C, Eich W, Harter M, Bieber C. Study protocol of a randomized controlled trial on two new dissemination strategies for a brief, shared-decision-making (SDM) training for oncologists: web-based interactive SDM online-training versus individualized context-based SDM face-to-face training. Trials. 2019 Jan 7;20(1):18. doi: 10.1186/s13063-018-3112-7. PMID 30616653
- See also: Study Homepage — http://www.pefmed.de